CLINICAL TRIAL: NCT01901419
Title: Nitroglycerin Infusion During Rewarming in Cardiac Surgery and Its Effects on Tissue Perfusion and Coagulation
Brief Title: Nitroglycerin Infusion During Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Tso-Chou Lin, MD, Assistant Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSGHIRB 1-102-05-049
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-10

CONDITIONS: Lactic Acidosis; Blood Glucose, High
Keywords: nitroglycerin; cardiopulmonary bypass; cardiac surgery
MeSH Terms: conditions — Acidosis, Lactic

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-dose NTG (Experimental): Nitroglycerin infusion 1-5 mcg/kg/min
  Interventions: Drug: Nitroglycerin infusion
- Low-dose NTG (Active Comparator): Nitroglycerin infusion 0-0.1 mcg/kg/min
  Interventions: Drug: Nitroglycerin infusion

INTERVENTIONS:
Drug: Nitroglycerin infusion — Nitroglycerin infusion during rewarming
  Other Names: Millisrol

SUMMARY:
Hypothermic cardiopulmonary bypass results in peripheral vasoconstriction and heparin trapping. Hypoperfusion and ischemic-reperfusion injury are associated with systemic inflammatory response, while insufficient and delayed neutralization of heparin by protamine may contribute to more blood loss during rewarming stage.

Nitroglycerin infusion, an NO-related vasodilator, is an established and effective treatment for unstable angina, myocardial infarction, congestive heart failure, and perioperative hemodynamic management for cardiac surgery. Therefore, we hypothesize that nitroglycerin infusion during rewarming corrects systemic ischemic stress and facilitates heparin neutralization in cardiac surgery.

DETAILED DESCRIPTION:
A randomized clinical trial in a tertiary academic center in patients with cardiac surgery, to receive either nitroglycerin infusion dose of 0-0.1 mcg/kg/min, or 1-5 mcg/kg/min during rewarming in cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery

Exclusion Criteria:

* heart failure, respiratory failure, asthma attack, uremia, normothermic bypass.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tso-Chou Lin, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication are to be shared starting 6 months after journal publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after journal publication.
Access Criteria: all IPD that underlie results in a publication are to be shared via email requests. The corresponding author will review requests and send them the supporting information.

REFERENCES:
- [Background] Piquette D, Deschamps A, Belisle S, Pellerin M, Levesque S, Tardif JC, Denault AY. Effect of intravenous nitroglycerin on cerebral saturation in high-risk cardiac surgery. Can J Anaesth. 2007 Sep;54(9):718-27. doi: 10.1007/BF03026868. PMID 17766739
- [Background] Masoumi G, Pour EH, Sadeghpour A, Ziayeefard M, Alavi M, Anbardan SJ, Shirani S. Effect of different dosages of nitroglycerin infusion on arterial blood gas tensions in patients undergoing on- pump coronary artery bypass graft surgery. J Res Med Sci. 2012 Feb;17(2):123-7. PMID 23264783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: elective cardiac surgery
Period: Overall Study
Arm/Group | High-dose NTG | Low-dose NTG
Started | 40 | 40
Completed | 32 | 31
Not Completed | 8 | 9
Not completed — Protocol Violation | 2 | 6
Not completed — unavailable researchers | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose NTG | Low-dose NTG | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: year] | 62.5 (12.2) | 59.3 (13.2) | 60.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 22 | 21 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 31 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 32 | 31 | 63
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 32 | 31 | 63
Plasma Lactate Level [Mean (Standard Deviation); unit: mmol/L] | 1.1 (0.5) | 1.0 (0.4) | 1.0 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Lactate Level, Before Incision
Description: Plasma Lactate Level, mmol/L, Before Incision
Time Frame: Before Incision
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mmol/L | 1.1 (0.5) | 1.0 (0.4)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.618, t-test, 2 sided

2. Primary Outcome: Plasma Lactate Level, Before Start of CPB
Description: Plasma Lactate Level, mmol/L, Before Start of CPB
Time Frame: Before Start of CPB
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mmol/L | 1.4 (0.7) | 1.6 (0.7)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.410, t-test, 2 sided

3. Primary Outcome: Plasma Lactate Level, Release of Aortic Clamp
Description: Plasma Lactate Level, mmol/L, Release of Aortic Clamp
Time Frame: Release of Aortic Clamp
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mmol/L | 3.1 (1.2) | 2.6 (1.0)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.088, t-test, 2 sided

4. Primary Outcome: Plasma Lactate Level, After Protamine Administration
Description: Plasma Lactate Level, mmol/L, After Cessation of CPB and Protamine Administration
Time Frame: After Protamine Administration
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mmol/L | 3.3 (1.2) | 3.0 (1.1)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.320, t-test, 2 sided

5. Primary Outcome: Plasma Lactate Level, Upon Arrival at ICU
Description: Plasma Lactate Level, mmol/L, Upon Arrival at ICU
Time Frame: Upon Arrival at ICU
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mmol/L | 3.4 (1.6) | 3.2 (1.5)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.512, t-test, 2 sided

6. Primary Outcome: Plasma Glucose Level, Before Incision
Description: Plasma Glucose Level, mg/dL, Before Incision
Time Frame: Before Incision
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mg/dL | 139.4 (47.4) | 124.2 (32.0)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.144, t-test, 2 sided

7. Primary Outcome: Plasma Glucose Level, Before Start of CPB
Description: Plasma Glucose Level, mg/dL, Before Start of CPB
Time Frame: Before Start of CPB
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mg/dL | 179.2 (62.3) | 165.7 (46.2)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.338, t-test, 2 sided

8. Primary Outcome: Plasma Glucose Level, Release of Aortic Clamp
Description: Plasma Glucose Level, mg/dL, Release of Aortic Clamp
Time Frame: Release of Aortic Clamp
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mg/dL | 174.5 (49.5) | 165.0 (29.3)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.356, t-test, 2 sided

9. Primary Outcome: Plasma Glucose Level, After Protamine Administration
Description: Plasma Glucose Level, mg/dL, After Cessation of CPB and Protamine Administration
Time Frame: After Protamine Administration
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mg/dL | 196.9 (53.8) | 205.7 (41.1)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.478, t-test, 2 sided

10. Primary Outcome: Plasma Glucose Level, Upon Arrival at ICU
Description: Plasma Glucose Level, mg/dL, Upon Arrival at ICU
Time Frame: Upon Arrival at ICU
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mg/dL | 206.4 (55.7) | 214.8 (46.3)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.515, t-test, 2 sided

11. Primary Outcome: Mean Arterial Blood Pressure ≤ 40 mmHg After Initiation of NTG Infusion
Description: Mean Arterial Blood Pressure ≤ 40 mmHg After Initiation of NTG Infusion During Rewarming of Cardiopulmonary Bypass
Time Frame: After Initiation of NTG infusion During Rewarming
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
Participants | 6 | 0
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p < 0.001, Fisher Exact

12. Secondary Outcome: Activated Coagulation Time, Before Start of CPB
Description: Activated Coagulation Time, sec, Before Start of CPB
Time Frame: Before Start of CPB
Measure: Mean (Standard Deviation); unit: second
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
second | 158.9 (19.8) | 153.1 (18.1)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.227, t-test, 2 sided

13. Secondary Outcome: Activated Coagulation Time, After Protamine Administration
Description: Activated Coagulation Time, sec, After Cessation of CPB and Protamine Administration
Time Frame: After Protamine Administration
Measure: Mean (Standard Deviation); unit: second
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
second | 144.2 (15.9) | 138.2 (15.3)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.141, t-test, 2 sided

14. Secondary Outcome: Post-op Dopamine Infusion
Description: Infusion Rate of Dopamine, mcg/kg/min, Upon Arrival at ICU
Time Frame: Upon Arrival at ICU
Measure: Mean (Standard Deviation); unit: mcg/kg/min
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
mcg/kg/min | 3.7 (1.8) | 4.7 (2.0)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.046, t-test, 2 sided

15. Secondary Outcome: Time to Extubation
Description: Time from Arrival at ICU to Extubation, hour
Time Frame: Arrival at ICU and Extubation
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
hour | 43.6 (33.7) | 45.8 (34.8)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.800, t-test, 2 sided

16. Secondary Outcome: Length of ICU Stay
Description: Time from Arrival at ICU to Leaving ICU, day
Time Frame: Arrival at ICU and Leaving ICU
Measure: Mean (Standard Deviation); unit: day
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
day | 4.1 (1.8) | 4.0 (2.0)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.948, t-test, 2 sided

17. Other Pre Specified Outcome: Cardiac Index, Before Start of CPB
Description: Cardiac Index, L/min/m2, Before Start of CPB
Time Frame: Before Start of CPB
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
L/min/m2 | 3.0 (1.3) | 2.8 (1.1)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.682, t-test, 2 sided

18. Other Pre Specified Outcome: Cardiac Index, Cessation of CPB
Description: Cardiac Index, L/min/m2, Cessation of CPB
Time Frame: Cessation of CPB
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
L/min/m2 | 2.6 (1.0) | 2.7 (0.6)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.928, t-test, 2 sided

19. Other Pre Specified Outcome: Cardiac Index, After Protamine Administration
Description: Cardiac Index, L/min/m2, After Protamine Administration
Time Frame: After Protamine Administration
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
L/min/m2 | 3.2 (1.0) | 3.1 (0.7)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.672, t-test, 2 sided

20. Other Pre Specified Outcome: Cardiac Index, Upon Arrival at ICU
Description: Cardiac Index, L/min/m2, Upon Arrival at ICU
Time Frame: Upon Arrival at ICU
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
L/min/m2 | 3.3 (0.9) | 3.3 (1.3)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.894, t-test, 2 sided

21. Other Pre Specified Outcome: Cerebral Oximetry, Before Start of CPB, Left Forehead
Description: Absolute Value of Cerebral Oximetry, %, Before Start of CPB, Left Forehead
Time Frame: Before Start of CPB
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 74.4 (4.8) | 76.8 (6.9)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.135, t-test, 2 sided

22. Other Pre Specified Outcome: Cerebral Oximetry, Before Start of CPB, Right Forehead
Description: Absolute Value of Cerebral Oximetry, %, Before Start of CPB, Right Forehead
Time Frame: Before Start of CPB
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 74.9 (4.6) | 77.9 (6.0)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.038, t-test, 2 sided

23. Other Pre Specified Outcome: Cerebral Oximetry, Beginning Rewarming, Left Forehead
Description: Absolute Value of Cerebral Oximetry, %, Beginning Rewarming, Left Forehead
Time Frame: Beginning Rewarming
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 68.0 (5.7) | 68.4 (7.8)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.852, t-test, 2 sided

24. Other Pre Specified Outcome: Cerebral Oximetry, Beginning Rewarming, Right Forehead
Description: Absolute Value of Cerebral Oximetry, %, Beginning Rewarming, Right Forehead
Time Frame: Beginning Rewarming
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 67.9 (7.2) | 69.5 (8.3)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.454, t-test, 2 sided

25. Other Pre Specified Outcome: Cerebral Oximetry, Release of Aortic Clamp, Left Forehead
Description: Absolute Value of Cerebral Oximetry, %, Release of Aortic Clamp, Left Forehead
Time Frame: Release of Aortic Clamp
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 67.4 (5.6) | 66.8 (5.8)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.663, t-test, 2 sided

26. Other Pre Specified Outcome: Cerebral Oximetry, Release of Aortic Clamp, Right Forehead
Description: Absolute Value of Cerebral Oximetry, %, Release of Aortic Clamp, Right Forehead
Time Frame: Release of Aortic Clamp
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 68.2 (6.1) | 67.9 (6.7)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.872, t-test, 2 sided

27. Other Pre Specified Outcome: Cerebral Oximetry, Cessation of CPB, Left Forehead
Description: Absolute Value of Cerebral Oximetry, %, Cessation of CPB, Left Forehead
Time Frame: Cessation of CPB
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 71.1 (4.0) | 69.8 (5.8)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.318, t-test, 2 sided

28. Other Pre Specified Outcome: Cerebral Oximetry, Cessation of CPB, Right Forehead
Description: Absolute Value of Cerebral Oximetry, %, Cessation of CPB, Right Forehead
Time Frame: Cessation of CPB
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 71.4 (4.9) | 70.0 (6.6)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.365, t-test, 2 sided

29. Other Pre Specified Outcome: Cerebral Oximetry, After Protamine Administration, Left Forehead
Description: Absolute Value of Cerebral Oximetry, %, After Protamine Administration, Left Forehead
Time Frame: After Protamine Administration
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 74.9 (4.3) | 72.1 (6.9)
Statistical Analysis 1: Comparison: High-dose NTG vs Low-dose NTG; Test type: Superiority; p = 0.077, t-test, 2 sided

30. Other Pre Specified Outcome: Cerebral Oximetry, After Protamine Administration, Right Forehead
Description: Absolute Value of Cerebral Oximetry, %, After Protamine Administration, Right Forehead
Time Frame: After Protamine Administration
Measure: Mean (Standard Deviation); unit: % of Cerebral Oximetry
Arm/Group | High-dose NTG | Low-dose NTG
Number analyzed (Participants) | 32 | 31
% of Cerebral Oximetry | 75.0 (4.7) | 74.3 (7.3)
Statistical Analysis 1: Comparison: High-dose NTG; Test type: Superiority; p = 0.640, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 30-day mortality and complications.
Description: Re-sternotomy for bleeding; Mediastinitis with septic shock; Pneumonia; Massive hemothorax
Arm/Group | High-dose NTG | Low-dose NTG
All-Cause Mortality (participants affected / at risk) | 1/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 2/32 | 2/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose NTG (N=32) | Low-dose NTG (N=31)
Re-sternotomy for bleeding (Surgical and medical procedures) | 1 (1) | 0 (0)
Mediastinitis with septic shock (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Massive hemothorax (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
One patient in NTG group experienced re-sternotomy to check bleeding in the same day and another one expired at the 25th day postoperatively due to mediastinitis with septic shock.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT01901419/Prot_SAP_000.pdf